CLINICAL TRIAL: NCT00433446
Title: A Phase II Study of CNTO 328, A Monoclonal Antibody Against Interleukin-6 (IL-6), in Patients With Hormone Refractory Prostate Cancer
Brief Title: S0354, Anti-IL-6 Chimeric Monoclonal Antibody in Patients With Metastatic Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000526555; U10CA032102 (NIH); S0354 (Other: SWOG)
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CNTO 328 (Experimental)
  Interventions: Biological: CNTO 328

INTERVENTIONS:
Biological: CNTO 328
  Other Names: anti-IL-6 chimeric monoclonal antibody

SUMMARY:
RATIONALE: Monoclonal antibodies, such as anti-IL-6 chimeric monoclonal antibody, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase II trial is studying how well anti-IL-6 chimeric monoclonal antibody works in treating patients with metastatic prostate cancer that did not respond to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the confirmed prostate-specific antigen response in patients with hormone-refractory metastatic prostate cancer treated with anti-IL-6 chimeric monoclonal antibody.

Secondary

* Assess overall survival and progression-free survival of these patients.
* Assess the objective response rate (confirmed and unconfirmed, complete and partial response) in patients with measurable disease treated with this regimen.
* Assess the qualitative and quantitative toxicities of this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive anti-IL-6 chimeric monoclonal antibody IV over 2 hours on day 1. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for up to 2 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Metastatic disease (N1 and/or M1)
* Disease unresponsive or refractory to androgen-deprivation therapy
* Must have received only 1 prior chemotherapy regimen comprising a taxane OR mitoxantrone
* Disease progression as defined by one or more of the following:

  * Progression of measurable disease

    * Prior radiotherapy allowed provided radiotherapy was completed ≥ 2 months ago and lesion progressed since radiotherapy
  * Progression of nonmeasurable disease

    * Prior radiotherapy within the past 2 months allowed, but disease is considered nonmeasurable
  * Rising prostate-specific antigen (PSA) after > 2 courses of chemotherapy OR within 6 months of last chemotherapy dose

    * Rising PSA defined as at least 2 consecutive rises in PSA to be documented over a reference value (measure 1)
* PSA ≥ 5 ng/mL
* Surgical or medical castration required

  * Castration using luteinizing hormone-releasing hormone agonist (leuprolide acetate or goserelin) or antagonist (abarelix) should not be interrupted
* No history of brain metastases OR currently treated or untreated brain metastases

  * Patients with clinical suspicion of brain metastases must have a brain CT scan or MRI negative for metastatic disease within the past 56 days

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Fertile patients must use effective contraception
* Absolute granulocyte count ≥ 1,500/mm³ (transfusion independent)
* Platelet count ≥ 100,000/mm³ (transfusion independent)
* Hemoglobin ≥ 9 g/dL (transfusion independent)
* Creatinine clearance ≥ 40 mL/min
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2 times ULN
* No uncontrolled intercurrent illnesses including, but not limited to, the following:

  * Diabetes mellitus
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No psychiatric illness or social situation that would preclude study compliance
* No known HIV positivity
* No other prior malignancy except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Adequately treated stage I or II cancer in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 21 days since prior surgery and recovered
* At least 28 days since prior chemotherapy and recovered
* At least 28 days since prior flutamide or ketoconazole
* At least 28 days since prior radiotherapy (to < 30% of the bone marrow only) and recovered

  * Prior samarium Sm 153 lexidronam pentasodium allowed
  * No prior strontium chloride Sr 89
* At least 42 days since prior bicalutamide or nilutamide
* More than 60 days since prior murine or chimeric proteins or human/murine monoclonal antibody
* Concurrent bisphosphonate therapy allowed provided the following are true:

  * Therapy commenced at least 3 weeks ago
  * Therapy continues for the entire duration of study treatment
* No other concurrent anticancer therapy, including cytotoxic therapy, biologic therapy, radiotherapy, or hormonal therapy (except for luteinizing hormone-releasing hormone agonist or antagonist in patients who have not had an orchiectomy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, MD, Study Chair — University of Southern California
Locations (123):
- United States (123):
  - Regional Medical Center, Anniston, Alabama
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Sutter Solano Medical Center, Vallejo, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Dorff TB, Goldman B, Pinski JK, Mack PC, Lara PN Jr, Van Veldhuizen PJ Jr, Quinn DI, Vogelzang NJ, Thompson IM Jr, Hussain MH. Clinical and correlative results of SWOG S0354: a phase II trial of CNTO328 (siltuximab), a monoclonal antibody against interleukin-6, in chemotherapy-pretreated patients with castration-resistant prostate cancer. Clin Cancer Res. 2010 Jun 1;16(11):3028-34. doi: 10.1158/1078-0432.CCR-09-3122. Epub 2010 May 18. PMID 20484019

RESULTS

PARTICIPANT FLOW:
Groups:
- CNTO 328: CNTO 328 will be given 6 mg/kg through intravenous (IV) once per cycle ( 1 cycle= 14 days) for 12 cycles
Period: Overall Study
Arm/Group | CNTO 328
Started | 62
Eligible | 53
Eligible and Began Protocol Therapy | 53
Completed | 1
Not Completed | 61
Not completed — Adverse Event | 4
Not completed — Refusal Unrelated to Adverse Event | 1
Not completed — Progression | 44
Not completed — Other - Not Protocol specified | 3
Not completed — Ineligible | 9

BASELINE CHARACTERISTICS:
Arm/Group | CNTO 328
Number analyzed (Participants) | 53
Age Continuous [Median (Full Range); unit: years] | 71 [46 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Baseline PSA (ng/dL) [Median (Full Range); unit: ng/dL] | 75.1 [6.3 to 10181]
Performance Status [Number; unit: participants] — Patients will be graded according to the Zubrod performance status scale. 0: Fully active, able to carry all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. 2: Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours. 3: Capable of limited self-care, confined to bed or chair more than 50% of waking hours. 4: Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  participants
    0 | 19
    1 | 28
    2 | 6
Prior Taxane Therapy [Number; unit: participants]
  Yes | 53
  No | 0

OUTCOME MEASURES:

1. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as tumor progression by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, PSA progression by PSA Working Group criteria, or symptomatic deterioration.
Time Frame: Assessed every 3 cycles (1 cycle = 14 days) until progression
Population: All eligible patients who started treatment were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CNTO 328
Number analyzed (Participants) | 53
months | 1.6 [1.6 to 1.7]

2. Primary Outcome: Confirmed Prostate-Specific Antigen (PSA) Response
Description: PSA response is defined as a 50% reduction in accordance with the recommendations of the orginal PSA Working Group. Confirmed PSA response is defined as PSA response at two or more time points at least 4 weeks apart, without objective disease progression or symptomatic deterioration.
Time Frame: Assessed every 3 cycles (1 cycle = 14 days) until progression
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CNTO 328
Number analyzed (Participants) | 53
percentage of participants | 3.8 [0.5 to 13.0]

3. Secondary Outcome: Overall Survival (OS)
Description: Measured from date of registration to date of death due to any cause or last contact
Time Frame: 0-3 yeas after registration
Population: All eligible patients who started treatment were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CNTO 328
Number analyzed (Participants) | 53
months | 11.6 [7.5 to 19]

4. Secondary Outcome: Objective Response (Confirmed and Unconfirmed Complete and Partial Response) Among Those Patients With Measurable Disease
Description: Complete Response (CR) is a complete disappearance of all measurable and non-measurable disease. No new lesions. No disease related symptoms. PSA = .2 ng/ml. Partial Response (PR) applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions.
Time Frame: Assessed every 3 cycles (1 cycle= 14 days) of treatment until progression
Population: All eligible patients with measurable disease who started treatment were included in the analysis
Measure: Number; unit: participants
Arm/Group | CNTO 328
Number analyzed (Participants) | 31
participants
  Complete Repsonse (CR) | 0
  Partial Response (PR) | 0
  Unconfirmed Complete Response | 0
  Unconfirmed Partial Response | 0
  Stable Disease | 7
  No response | 24

5. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Patients were assessed for adverse events after every cycle (1 cycle = 14 days) of protocol treatment
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | CNTO 328
Number analyzed (Participants) | 53
Participants
  AST, SGOT | 1
  Alkaline phosphatase | 1
  CNS cerebrovascular ischemia | 1
  DIC (disseminated intravascular coagulation) | 1
  Esophagitis | 1
  Gastritis (including bile reflux gastritis) | 1
  Leukocytes (total WBC) | 1
  Neuropathy: motor | 1
  Neutrophils/granulocytes (ANC/AGC) | 1
  Pain - Muscle | 1
  Pain-Other (Specify: hip and back) | 1
  Platelets | 2

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events after every cycle (1 cycle = 14 days) of protocol treatment
Arm/Group | CNTO 328
Serious Adverse Events (participants affected / at risk) | 9/53
Other Adverse Events (participants affected / at risk) | 47/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CNTO 328 (N=53)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1
Extremity-lower (gait/walking) (General disorders) | 1
Sudden death (General disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Stricture/stenosis (incl anastomotic), GU - Ureter (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hematoma (Vascular disorders) | 1
Vascular-Other (Specify) (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CNTO 328 (N=53)
Hemoglobin (Blood and lymphatic system disorders) | 18
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 22
Pain - Abdomen NOS (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 10
Edema: limb (General disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 28
Pain-Other (Specify) (General disorders) | 7
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4
AST, SGOT (Investigations) | 10
Alkaline phosphatase (Investigations) | 11
Bilirubin (hyperbilirubinemia) (Investigations) | 3
INR (of prothrombin time) (Investigations) | 3
Leukocytes (total WBC) (Investigations) | 15
Lymphopenia (Investigations) | 7
Metabolic/Laboratory-Other (Specify) (Investigations) | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6
Platelets (Investigations) | 9
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 8
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13
Pain - Back (Musculoskeletal and connective tissue disorders) | 12
Pain - Bone (Musculoskeletal and connective tissue disorders) | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 5
Pain - Joint (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 9
Neuropathy: sensory (Nervous system disorders) | 11
Pain - Head/headache (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 5
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 3
Erectile dysfunction (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Hot flashes/flushes (Vascular disorders) | 4
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No